CLINICAL TRIAL: NCT02134821
Title: Influence of Pain Sensitivity on Surgical Outcomes After Lumbar Spine Surgery in Patients With Lumbar Spinal Stenosis
Brief Title: Influence of Pain Sensitivity on Lumbar Surgery Outcomes
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Other Study IDs: PSQ_001
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Low pain sensitivity group: total Pain Sensitivity Questionnaire score <6.5
  Interventions: Procedure: Surgery for lumbar spinal stenosis
- High pain sensitivity group: total pain sensitivity questionnaire score ≥ 6.5
  Interventions: Procedure: Surgery for lumbar spinal stenosis

INTERVENTIONS:
Procedure: Surgery for lumbar spinal stenosis — decompression with or without fusion for lumbar spinal stenosis

SUMMARY:
Pain sensitivity would be associated with surgical outcomes after lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 40-80 years
2. lumbar spinal stenosis diagnosis and scheduled spine surgery at a tertiary-care teaching institution between June 2012 and April 2013

Exclusion Criteria:

* a history of major psychiatric disorders (schizophrenia, major depression) or peripheral vascular disease
* any concurrent serious medical condition that would cause disability or decreased general health status such as sepsis or cancer.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria were the following: 1) patients aged 40-80 years; 2) an lumbar spinal stenosis diagnosis and scheduled spine surgery at a tertiary-care teaching institution between June 2012 and April 2013
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | up to 12 months after operation

SECONDARY OUTCOMES:
Visual Analog Pain Scale for back pain | up to 12 months after operation
Visual Analog Pain Scale for leg pain | up to 12 months after operation
Short-Form 36 | up to 12 months after operation
  measurement of general health status

CONTACTS AND LOCATIONS:
Overall Officials: Jin S. Yeom, MD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Sung-Nam, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim HJ, Park JW, Kang KT, Chang BS, Lee CK, Kang SS, Yeom JS. Determination of the Optimal Cutoff Values for Pain Sensitivity Questionnaire Scores and the Oswestry Disability Index for Favorable Surgical Outcomes in Subjects With Lumbar Spinal Stenosis. Spine (Phila Pa 1976). 2015 Oct 15;40(20):E1110-6. doi: 10.1097/BRS.0000000000001023. PMID 26076437